CLINICAL TRIAL: NCT04633226
Title: A Phase 3, Single-Arm, Open-label Clinical Study to Evaluate the Safety and Immunogenicity of 4 Doses of V114 Administered to Healthy Infants in South Korea.
Brief Title: Safety and Immunogenicity of V114 in Healthy Infants in South Korea (V114-036)
Acronym: PNEU-PED-KOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V114-036; V114-036 (Other: MSD); 2020-003181-39 (EudraCT Number)
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V114 (Experimental): Participants received 4 total doses of V114, administered at approximately 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114

INTERVENTIONS:
Biological: V114 — 15-valent pneumococcal conjugate vaccine (PCV) containing 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) present in Prevnar 13™ plus 2 additional serotypes (22F, 33F) in each 0.5 mL sterile suspension for intramuscular injection.
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine

SUMMARY:
The primary purpose of this phase 3, single-arm, open-label study is to evaluate the safety and immunogenicity of a 4-dose regimen of V114 administered to healthy infants in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* is a healthy South Korean male or female who is 42 to 90 days of age at the time of signing informed consent
* has a parent or legally acceptable representative who understands study procedures, alternative treatments available, and risks involved and voluntarily agrees to participate by signing informed consent

Exclusion Criteria:

* has a history of invasive pneumococcal disease or known history of other culture positive pneumococcal disease
* has known hypersensitivity to pneumococcal conjugate vaccine, any licensed pediatric vaccine to be administered concomitantly, or any diphtheria toxoid-containing vaccine
* has had a recent febrile illness (rectal temperature ≥38.1°C [≥100.5°F] or axillary temperature ≥37.8°C [≥100.0°F]) within 72 hours prior to receipt of study vaccine
* has known or suspected impairment of immunological function
* has or his/her mother has human immunodeficiency virus (HIV) infection
* has or his/her mother has hepatitis B surface antigen-positive test
* has known or history of functional or anatomic asplenia
* has a history of autoimmune disease
* has a history or suspected history of neurological disorder
* has received a pneumococcal vaccine prior to study entry
* has received, or is anticipated to need, corticosteroid therapy
* has received a blood transfusion of immunoglobulin products
* has participated in another clinical study of an investigational product

Ages: 42 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (19):
- South Korea (19):
  - Jeonbuk National University Hospital ( Site 0008), Jeonju, Jeonrabugdo
  - Korea University Ansan Hospital ( Site 0006), Ansan-si, Kyonggi-do
  - Hallym University Sacred Heart Hospital ( Site 0011), Anyang-si, Kyonggi-do
  - Hallym University Dongtan Sacred Heart Hospital ( Site 0013), Hwaseong-si, Kyonggi-do
  - CHA Bundang Medical Center CHA University ( Site 0020), Seongnam-si, Kyonggi-do
  - Changwon Fatima Hospital ( Site 0015), Changwon, Kyongsangnam-do
  - Pusan National University Yangsan Hospital ( Site 0009), Yangsan, Kyongsangnam-do
  - Kyungpook National University Hospital ( Site 0014), Daegu, Taegu-Kwangyokshi
  - The Catholic University of Korea, Incheon St. Mary's Hospital ( Site 0012), Incheon
  - Gachon University Gil Medical Center ( Site 0019), Incheon
  - Inha University Hospital ( Site 0001), Incheon
  - Korea Cancer Center Hospital ( Site 0017), Seoul
  - Nowon Eulji Medical Center, Eulji University ( Site 0005), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0002), Seoul
  - Samsung Medical Center ( Site 0007), Seoul
  - The Catholic University of Korea ( Site 0003), Seoul
  - Chung-Ang University Hospital ( Site 0016), Seoul
  - Ewha Womans University Seoul Hospital ( Site 0010), Seoul
  - Korea University Guro Hospital ( Site 0021), Seoul

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Maestri A, Park SE, Fernandes F, Li ZL, Kim YJ, Kim YK, Lee J, Park JY, Kim DH, Yang G, Lim H, Kim JO, Lupinacci R, Sterling TM, Wilck M, Esteves-Jaramillo A, Banniettis N. A phase 3, single-arm, open-label study to evaluate the safety, tolerability, and immunogenicity of a 15-valent pneumococcal conjugate vaccine, V114, in a 3+1 regimen in healthy infants in South Korea (PNEU-PED-KOR). Hum Vaccin Immunother. 2024 Dec 31;20(1):2321035. doi: 10.1080/21645515.2024.2321035. Epub 2024 Mar 18. PMID 38497448
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26088&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | V114
Started | 58
Vaccination 1 (~2 Months of Age) | 57
Vaccination 2 (~4 Months of Age) | 56
Vaccination 3 (~6 Months of Age) | 55
Vaccination 4 (~12 to 15 Months of Age) | 50
Completed | 53
Not Completed | 5
Not completed — Withdrawal by parent/guardian | 4
Not completed — Randomized by mistake without study treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | V114
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 8.7 (1.2)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0
  Preterm newborn infants (gestational age < 37 wks) | 0
  Newborns (0-27 days) | 0
  Infants and toddlers (28 days-23 months) | 58
  Children (2-11 years) | 0
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 0
  From 65-84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 58
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥1 Solicited Injection-site Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following any of the doses of V114, the percentage of participants with solicited injection-site AEs was assessed. The solicited injection-site AEs consist of erythema, induration, pain, and swelling.
Time Frame: Up to 7 days after any vaccination, up to a total of ~ 13 months
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114
Number analyzed (Participants) | 57
Percentage of Participants
  Injection site erythema | 54.4
  Injection site induration | 57.9
  Injection site pain | 50.9
  Injection site swelling | 59.6

2. Primary Outcome: Percentage of Participants With ≥1 Solicited Systemic Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following any of the doses of V114, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs consist of decreased appetite, irritability, somnolence, and urticaria.
Time Frame: Up to 7 days after any vaccination, up to a total of ~ 13 months
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114
Number analyzed (Participants) | 57
Percentage of Participants
  Decreased appetite | 71.9
  Irritability | 89.5
  Somnolence | 82.5
  Urticaria | 8.8

3. Primary Outcome: Percentage of Participants With ≥1 Vaccine-related Serious Adverse Events
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants with a vaccine-related SAE following any dose of V114 was reported. Vaccine-related SAEs were counted starting after vaccine dose 1 through completion of study.
Time Frame: Up to approximately 14.5 months
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114
Number analyzed (Participants) | 57
Percentage of Participants | 0.0 (0.0) [0.0 to 6.3]

4. Primary Outcome: Percentage of Participants Discontinuing Study Therapy Due to an Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The percentage of participants who discontinued study treatment due to an AE is reported.
Time Frame: Up to approximately 13 months
Population: The analysis population consisted of all participants who received at least 1 dose of study vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114
Number analyzed (Participants) | 57
Percentage of Participants | 0.0 (0.0) [0.0 to 6.3]

5. Primary Outcome: Percentage of Participants With Anti-Pneumococcal Polysaccharides Serotype-specific Immunoglobulin G ≥0.35 µg/mL
Description: The percentage of participants with immunoglobulin G (IgG) threshold values of ≥0.35 µg/mL for the 15 serotypes contained in V114 (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F) at 30 days postdose 3 is reported. The multiplex, pneumococcal electrochemiluminescence (PnECL) v2.0 assay was used to quantify IgG serotype-specific antibodies.
Time Frame: 30 days after vaccination 3 (Up to a total of ~5 months)
Population: All randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity endpoint and who had sufficient data to perform the analyses were analyzed. Deviations include randomized but not vaccinated, prior pneumococcal vaccine, vaccination out of window, blood draw out of window, prohibited concomitant medication or vaccine, or missing serology results.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114
Number analyzed (Participants) | 47
Percentage of Participants
  Serotype 1 | 100.0 [92.5 to 100.0]
  Serotype 3 | 100.0 [92.5 to 100.0]
  Serotype 4 | 100.0 [92.5 to 100.0]
  Serotype 5 | 100.0 [92.5 to 100.0]
  Serotype 6A | 100.0 [92.5 to 100.0]
  Serotype 6B | 95.7 [85.5 to 99.5]
  Serotype 7F | 100.0 [92.5 to 100.0]
  Serotype 9V | 100.0 [92.5 to 100.0]
  Serotype 14 | 100.0 [92.5 to 100.0]
  Serotype 18C | 97.9 [88.7 to 99.9]
  Serotype 19A | 97.9 [88.7 to 99.9]
  Serotype 19F | 100.0 [92.5 to 100.0]
  Serotype 22F | 100.0 [92.5 to 100.0]
  Serotype 23F | 100.0 [92.5 to 100.0]
  Serotype 33F | 97.9 [88.7 to 99.9]

6. Primary Outcome: Geometric Mean Concentrations of Anti-Pneumococcal Polysaccharides Serotype-specific Immunoglobulin G at 30 Days Postdose 3
Description: The anti-pneumococcal polysaccharides (PnPs) serotype-specific IgG geometric mean concentrations (GMCs) at 30 days postdose 3 for each serotype-specific were reported. The multiplex, electrochemiluminescence (ECL)-based PnECL v2.0 assay was used to quantify IgG serotype-specific antibodies.
Time Frame: 30 days after vaccination 3 (Up to a total of ~5 months)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114
Number analyzed (Participants) | 47
μg/mL
  Serotype 1 | 1.69 [1.46 to 1.94]
  Serotype 3 | 1.70 [1.41 to 2.06]
  Serotype 4 | 1.87 [1.49 to 2.34]
  Serotype 5 | 2.14 [1.74 to 2.63]
  Serotype 6A | 2.16 [1.74 to 2.67]
  Serotype 6B | 2.53 [1.93 to 3.32]
  Serotype 7F | 2.80 [2.35 to 3.32]
  Serotype 9V | 2.01 [1.63 to 2.47]
  Serotype 14 | 7.47 [5.98 to 9.32]
  Serotype 18C | 1.90 [1.47 to 2.46]
  Serotype 19A | 2.20 [1.76 to 2.76]
  Serotype 19F | 3.04 [2.55 to 3.63]
  Serotype 22F | 5.97 [4.83 to 7.37]
  Serotype 23F | 1.71 [1.37 to 2.15]
  Serotype 33F | 2.41 [1.84 to 3.15]

7. Secondary Outcome: Geometric Mean Concentrations of Anti-Pneumococcal Polysaccharides Serotype-specific Immunoglobulin G at 30 Days Postdose 4
Description: The anti-PnPs serotype-specific IgG GMCs at 30 days postdose 4 for each serotype-specific were reported. The multiplex, ECL-based PnECL v2.0 assay was used.
Time Frame: 30 days after vaccination 4 (Up to a total of ~14 months)
Population: All randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity endpoint and who had sufficient data to perform the analyses were analyzed. Deviations include vaccination out of window, blood draw out of window, or prohibited concomitant medication or vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114
Number analyzed (Participants) | 49
μg/mL
  Serotype 1 | 2.24 [1.77 to 2.83]
  Serotype 3 | 1.32 [1.07 to 1.62]
  Serotype 4 | 1.86 [1.39 to 2.49]
  Serotype 5 | 3.27 [2.57 to 4.17]
  Serotype 6A | 5.77 [4.38 to 7.60]
  Serotype 6B | 6.80 [5.28 to 8.76]
  Serotype 7F | 5.17 [3.92 to 6.81]
  Serotype 9V | 3.27 [2.50 to 4.28]
  Serotype 14 | 9.04 [7.22 to 11.31]
  Serotype 18C | 3.81 [2.97 to 4.88]
  Serotype 19A | 4.91 [4.03 to 5.97]
  Serotype 19F | 5.41 [4.40 to 6.65]
  Serotype 22F | 9.20 [7.19 to 11.79]
  Serotype 23F | 2.82 [2.14 to 3.73]
  Serotype 33F | 6.21 [5.05 to 7.63]

ADVERSE EVENTS:
Time Frame: Up to ~14.5 months
Description: All-Cause Mortality was reported for all allocated participants. The analysis population for AEs included all allocated participants who received at least 1 dose of study treatment.
Arm/Group | V114
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 4/57
Other Adverse Events (participants affected / at risk) | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=57)
Pyrexia (General disorders) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=57)
Diarrhoea (Gastrointestinal disorders) | 3 (5)
Injection site erythema (General disorders) | 31 (64)
Injection site induration (General disorders) | 33 (70)
Injection site pain (General disorders) | 29 (73)
Injection site swelling (General disorders) | 34 (72)
Injection site urticaria (General disorders) | 9 (13)
Pyrexia (General disorders) | 19 (27)
Nasopharyngitis (Infections and infestations) | 5 (7)
Decreased appetite (Metabolism and nutrition disorders) | 41 (65)
Somnolence (Nervous system disorders) | 47 (108)
Irritability (Psychiatric disorders) | 51 (138)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT04633226/Prot_SAP_000.pdf